CLINICAL TRIAL: NCT01851746
Title: A Study of Docetaxel and Lobaplatin vs. Docetaxel and Carboplatin Combination Regimen in Patients With Platinum-sensitive (>6 Months) Relapsed Ovarian Cancer
Brief Title: A Study of Docetaxel and Lobaplatin Versus Docetaxel and Carboplatin Combination Regimen in Patients With Platinum-sensitive (>6 Months) Relapsed Ovarian Cancer
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Wuhan University (Other)
Responsible Party: Principal Investigator, HB Cai, Director of gynecologic oncology department of Zhongnan Hospital of Wuhan University, Wuhan University
Other Study IDs: CHB2013
Record Dates: First submitted 2013-05-07; First posted 2013-05-10 (Estimated); Last update posted 2013-05-10 (Estimated); Status verified 2013-05

CONDITIONS: Recurrent Ovarian Cancer
Keywords: recurrent ovarian cancer; lobaplatin; docetaxel; carboplatin
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Boold,Urine
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to evaluate the effectiveness and security of lobaplatin combined with docetaxel in treatment of the sensitive recurrent ovarian cancer.

ELIGIBILITY:
Inclusion Criteria:

1. age between 18 and 70 years old
2. singed the information consent form
3. Expected survival time >3 months
4. Recurrence for at least 6 months after receiving initial platinum-based chemotherapy and without cytoreductive surgery indications.

Exclusion Criteria:

1. Recurrence within 6 months after receiving initial platinum-based chemotherapy
2. without radiographic evidence for tumor recurrence
3. receiving other chemotherapy, hormone therapy, immunotherapy, or radiation therapy

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: residents of a certain town
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2013-03; Primary Completion 2015-02 (Estimated); Study Completion 2015-02 (Estimated)

PRIMARY OUTCOMES:
Evidence of the effectiveness and security of lobaplatin combined with docetaxel in treatment of the sensitive recurrent ovarian cancer. | from pre-chemotherapy to 4-6 weeks post-chemotherapy
  Blood routine, urine routine, hepatic and kidney function, electrolyte, ECG, CT,MRI

CONTACTS AND LOCATIONS:
Overall Officials: Hong-bing Cai, MD,PhD, Study Director — Zhongnan Hospital
Locations (1):
- Zhongnan Hospital of Wuhan University, Wuhan, Hubei, China